CLINICAL TRIAL: NCT06822413
Title: A Novel Raman Spectroscopy-Based Method for Pan-Cancers Early Diagnosis Supported by Deep Learning: A Prospective, Single-Arm, Multicentre Study
Brief Title: Raman Spectroscopy-Based Deep Learning Model for Early Pan-Cancer Early Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: The First Affiliated Hospital of Nanchang University (Other); Second Affiliated Hospital of Nanchang University (Other); Huashan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1060
Record Dates: First submitted 2025-02-05; First posted 2025-02-12 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-01

CONDITIONS: Cancer Diagnosis; Liver Cancer, Adult; Cancer Screening; Colorectal Cancer (CRC); Gastric Cancers; Normal Physiology; Pancreatic Cancer, Adult; Raman Spectroscopy; Deep Learning Model; Esophageal Cancer; Malignant Tumours; Precancerous Conditions; Pancreatitis; Adenoma Colon Polyp; Gastric Ulcer; Oesophagitis; Cirrhoses, Liver
Keywords: Pan-cancer; Deep Learning Models; Cancer Screening; Raman Spectroscopy; Colorectal Cancer; Pancreatic Cancer; Gastric Cancer; Esophageal Cancer; malignant tumour; Precancerous Condtions; Pancreatitis; Colorectal Adenoma; Gastirc Ulcer; Oesophagitis; Cirrhoses
MeSH Terms: conditions — Carcinoma, Hepatocellular; Colorectal Neoplasms; Stomach Neoplasms; Pancreatic cancer, adult; Esophageal Neoplasms; Neoplasms; Precancerous Conditions; Pancreatitis; Stomach Ulcer; Esophagitis; Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (11):
- Normal Physiology: Patients without cancers or precancerous lesion
  Interventions: Other: No Interventions
- Colorectal Cancer: Patients diagnosed with colorectal cancer (Pre-intervention)
  Interventions: Other: No Interventions
- Gastric Cancer: Patients diagnosed with gastric cancer (Pre-intervention)
  Interventions: Other: No Interventions
- Hepatic Cancer: Patients diagnosed with hepatic cancer (Pre-intervention)
  Interventions: Other: No Interventions
- Oesophageal: Patients diagnosed with oesophageal cancer (Pre-intervention)
- Pancreatic Cancer: Patients diagnosed with pancreatic cancer (Pre-intervention)
  Interventions: Other: No Interventions
- Gastric Ulcer: Patients with gastric ulcers without any cancer
  Interventions: Other: No Interventions
- Colorectal Adenoma: Patients with colorectal adenoma without any cancer
  Interventions: Other: No Interventions
- Liver Cirrhosis: Patients with liver cirrhosis without any cancer
  Interventions: Other: No Interventions
- Pancreatitis: Patients with pancreatitis without any cancer
  Interventions: Other: No Interventions
- Oesophagitis: Patients with oesophagitis without any cancer
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — All blood samples from participating patients were obtained from routine clinical blood tests conducted during hospital admission or other necessary medical evaluations, followed by serum extraction.
  Groups: Colorectal Adenoma; Colorectal Cancer; Gastric Cancer; Gastric Ulcer; Hepatic Cancer; Liver Cirrhosis; Normal Physiology; Oesophagitis; Pancreatic Cancer; Pancreatitis

SUMMARY:
The goal of this observational study is to explore whether a Raman-based, deep learning-assisted approach can be used to develop an effective method for early pan-cancer screening. The study includes healthy individuals, patients at risk of cancer, and patients with diagnosed cancers. The main questions it aims to answer are:

* Evaluating the deep-learning model's accuracy and specificity in identifying cancer-specific features in Raman spectral data and determining whether this method can accurately classify patients based on risk.
* Identifying which model is more adaptable to the Raman spectrum
* Providing an interpretable analysis of the model-generated diagnosis Participants are already being diagnosed and follow-up to determine the type of cancer.

DETAILED DESCRIPTION:
This study aims to explore the use of deep learning models for classifying patients based on Raman spectroscopy analysis of blood samples, distinguishing between individuals in physiological conditions and patients with various types of precancerous conditions or malignant tumors. The study is conducted through a multi-center collaboration, where blood samples are collected from both healthy participants and patients with histopathologically diagnosed precancerous conditions or primary malignant tumors.

All blood samples are obtained from patients' routine clinical blood tests conducted during hospital admission or other necessary medical evaluations. The spectral data undergo a rigorous preprocessing pipeline, which includes alignment resampling to standardize the data, baseline removal to eliminate unwanted variations, and normalization to ensure uniformity across all samples. The data is optimized for deep learning model training.

Various deep-learning models are then employed to analyze the processed Raman spectra and develop a classification system to distinguish between pan-cancer cases and healthy controls. The preprocessed dataset is partitioned into three subsets for model training and performance evaluation: 80% for training, 10% for validation, and 10% for testing. These datasets are used for model training to identify patterns in the spectral data that correlate with the presence of specific cancers or a healthy state, enabling accurate classification.

To enhance the interpretability of deep learning models, Grad-CAM (Gradient-weighted Class Activation Mapping) is used to visualize the models' decision-making processes. This allows the identification of the Raman spectra regions that are more influential in the model's classification decision, providing a transparent understanding of how the model differentiates between the various classes.

Ultimately, this study aims to demonstrate the potential of Raman spectroscopy combined with deep learning techniques as a non-invasive, accurate, and interpretable method for cancer detection and classification, with implications for early diagnosis and personalized treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Histopathological diagnosis of malignant tumors, including colorectal cancer, gastric cancer, hepatic cancer, pancreatic cancer, and esophageal cancer.
* Patients in normal physiological conditions without any malignant tumors or precancerous lesions.
* Patients with malignant tumor without recieving any interventions, including chemotherapy, surgery, radiotherapy, immunotherapy or other anti-tumor treatments.
* Patients with a histopathological diagnosis of any precancerous lesions or non-malignant disease.

Exclusion Criteria:

* Patients with metastatic tumors or in the condition with two or more kinds of malignant tumors at the same time
* Post-cancer treatment patients.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pan-cancer patients from Zhejiang, Jiangxi and Shanghai province
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-07-28 (Estimated)

PRIMARY OUTCOMES:
A Deep Learning Model for High-Accuracy Pan-Cancer Classification | From patient enrollment to the completion of model construction, expected to be finalized within two months after data collection.
  Establish deep learning models with high specificity and sensitivity for pan-cancer classification, capable of distinguishing different pan-cancer types (Distinguish between patients in physiological conditions, precancerous lesion and malignant tumour) based on Raman spectroscopy.

SECONDARY OUTCOMES:
Raman Shift Characteristics for Model Decision Interpretation and Visualization | From the end of model construction to the end of model interpretable analysis - expected 2 months after model construction
  Performing interpretable analysis of the diagnosis derived from the primary outcome using Grad-CAM to visualize and illustrate the model's decision-making process.

CONTACTS AND LOCATIONS:
Overall Officials: Kefeng Ding, MD, Study Chair — Department of Colorectal Surgery, The Second Hospital of Zhejiang University School of Medicine
Locations (4):
- China (4):
  - The First Affiliated Hospital to Nanchang University, Nanchang, Jiangxi
  - The Second Affiliated Hospital to Nanchang University, Nanchang, Jiangxi
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No